CLINICAL TRIAL: NCT03829475
Title: A Randomized Controlled Trial to Compare the Effectiveness of Fecal Microbiota Transplantation (FMT) in Combination With Bezlotoxumab Compared to FMT and Placebo for the Prevention of CDI Recurrence in Patients With Inflammatory Bowel Disease and Recurrent Clostridium Difficile Infection
Brief Title: ICON-2: FMT and Bezlotoxumab Compared to FMT and Placebo for Patients With IBD and CDI
Acronym: ICON-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jessica Ravikoff Allegretti, Director, Fecal Microbiota Transplantation Program, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018
Record Dates: First submitted 2019-01-26; First posted 2019-02-04 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Inflammatory Bowel Diseases; Clostridium Difficile Infection
Keywords: Crohn's DIsease; Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Clostridium Infections; Crohn Disease; Colitis, Ulcerative | interventions — bezlotoxumab; Sodium Chloride; Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FMT + Bezlo (Experimental): Patients in this arm will received an FMT via colonoscopy ( 250ml) as well as a single IV infusion of bezlotoxumab (10mg/kg) that will take place over 60 mins.
  Interventions: Drug: Bezlotoxumab; Drug: Fecal Microbiota Transplantation
- FMT + Placebo (Placebo Comparator): Patients in this arm will receive a single FMT via colonoscopy (250ml) and a placebo (saline) infusion (250cc) over
  Interventions: Drug: Placebo; Drug: Fecal Microbiota Transplantation

INTERVENTIONS:
Drug: Bezlotoxumab — This is a a fully human monoclonal antibody that binds to C. difficile toxin B, and is indicated to prevent recurrence of CDI in adults at risk for recurrent CDI (rCDI).
  Other Names: Zinplava
  Arms: FMT + Bezlo
Drug: Placebo — placebo is an infusion of normal saline.
  Other Names: Saline
  Arms: FMT + Placebo
Drug: Fecal Microbiota Transplantation — FMT is an infusion of prescreened donor stool that will be administered via colonoscopy
  Other Names: FMT

SUMMARY:
This is a randomized controlled trial to assess the clinical and microbiological impacts of FMT in combination with Bezlotoxumab (bezlo) compared to FMT in combination with placebo in patients with both inflammatory bowel disease (IBD) a and clostridium difficile infection (CDI). The investigators will prospectively enroll up to 150 IBD-CDI patients from 4 tertiary care FMT referral centers. Patients will be randomized 1:1 to either receive FMT in combination with Bezlo of FMT and a placebo infusion. Donor stool from healthy donors will be obtained from OpenBiome. OpenBiome is a nonprofit 501(c)(3) organization that provides hospitals with screened, filtered, and frozen material ready for clinical use. Patients will be enrolled and followed prospectively for 3 months post therapy. Stool and blood samples as well as clinical data will be collected at baseline, week 1, 8 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 or greater
* History of ≥ 2 episodes of recurrent CDI. CDI is defined as the presence of diarrhea ( Bristol 6 or 7 for 48 hours and a confirmatory test for CDI). Preferred testing will be a two-step method using GDH/EIA toxin, though PCR will be accepted based on hospital availability with confirmation of the most recent episode occurring within the prior 3 months
* Confirmed diagnosis of IBD (ulcerative colitis, Crohn's disease or indeterminate colitis)
* Undergoing FMT via colonoscopy for CDI as part of standard medical care

Exclusion Criteria:

* Unable or unwilling to undergo a colonoscopy
* Inpatient status, though patients can be screened while inpatients, the must be outpatient for the planned colonoscopy.
* Anticipated immediate or upcoming surgery within 30 days
* Need for continued non-anti-CDI antibiotic therapy
* History of total proctocolectomy
* Female patients who are pregnant or breastfeeding or plan to become pregnant in the next 6 months.
* Patients who are unable to give informed consent
* Participation in a clinical trial in the preceding 30 days or simultaneously during this trial
* Severe food allergy (anaphylaxis or anaphylactoid-like reaction)
* Life expectancy < 6 months
* Unable to adhere to protocol requirements
* Patient who have received an FMT in the past year
* Any condition that the physician investigators deems unsafe, including other conditions or medications that the investigator determines that it will put the subject at greater risk from FMT
* Patient who is diagnosed with NYHA class 3 or 4 Heart Failure
* Lab value of WBC <3.0 x 103/mm3 , Platelets <100 x 103/mm3 , ALT or AST > 1.5 x institutional ULN
* EBV or CMV negative if a patient is severely immunosuppressed ( defined as 3 or more immunosuppressing agents)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2025-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- FMT + Bezlo: Participants received an FMT via colonoscopy (250ml) as well as a single IV infusion of bezlotoxumab (10mg/kg) that took place over 60 minutes.
  Bezlotoxumab: This is a a fully human monoclonal antibody that binds to C. difficile toxin B, and is indicated to prevent recurrence of CDI in adults at risk for recurrent CDI (rCDI).
  Fecal Microbiota Transplantation: FMT is an infusion of prescreened donor stool that will be administered via colonoscopy
- FMT + Placebo: Participants received a single FMT via colonoscopy (250ml) and a placebo (saline) infusion (250cc) over 60 minutes.
  Placebo: placebo is an infusion of normal saline.
  Fecal Microbiota Transplantation: FMT is an infusion of prescreened donor stool that will be administered via colonoscopy
Period: Overall Study
Arm/Group | FMT + Bezlo | FMT + Placebo
Started | 30 | 31
Completed | 30 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FMT + Bezlo | FMT + Placebo | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38.5 [29 to 60] | 34 [28 to 54] | 38 [28 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 16 | 17 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 27 | 27 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Baseline Calprotectin [Median (Inter-Quartile Range); unit: mcg/g] | 930.5 [241 to 2950] | 241 [100 to 1615] | 635 [150 to 2615]
Baseline Bowel Movement [Median (Inter-Quartile Range); unit: bowel movements] — This is based on symptoms experienced in the 3 days preceding the baseline study visit.
  bowel movements | 5 [3 to 10] | 4 [3 to 6] | 5 [3 to 8]
Baseline Bristol Score [Median (Inter-Quartile Range); unit: units on a scale] — Range 1-7. Low scores represent hard stools and high numbers represent liquid stools
  units on a scale | 5 [4 to 6] | 5 [4 to 6] | 5 [4 to 6]
Baseline Partial Mayo [Median (Inter-Quartile Range); unit: units on a scale] — Range 0-9. The score is a ulcerative colitis disease activity assessment and has 3 components: bowel movements, rectal bleeding, and physical global assessment. Each component ranges from 0-3. The scores from each subsection are added together to get the total score. Low scores indicate inactive disease. High scores indicate active disease. Population: Partial Mayo only applies to subjects with Ulcerative Colitis
  units on a scale
    number analyzed (Participants) | 24 | 17 | 41
    (all) | 3.5 [2 to 5.5] | 2 [0 to 4] | 3 [2 to 5]
Baseline Harvey Bradshaw Index [Median (Inter-Quartile Range); unit: units on a scale] — This is a disease activity index for Crohn's disease. Components include: general well being [score 0-4] abdominal pain [score 0-3], number of liquid stools, abdominal mass [score 0-3], and complications of disease [score 0-8]. The score if each component is added together to get the total score [Range 0 to 18] The upper range is open ended as the number of liquid stools will vary by patient. HBI < 5 is defined as clinical remission, HBI between 5 and 7 as mild disease, HBI between 8 and 16 as moderate disease, and HBI > 16 as severe disease. Population: HBI only applies to subjects with Crohn's Disease
  units on a scale
    number analyzed (Participants) | 6 | 14 | 20
    (all) | 7 [2 to 11] | 6.5 [3 to 11] | 6.5 [3 to 11]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clostridium Difficile Recurrence
Description: positive test for CDI by EIA toxin
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | FMT + Bezlo | FMT + Placebo
Number analyzed (Participants) | 30 | 31
Participants | 4 | 1
Statistical Analysis 1: Comparison: FMT + Bezlo vs FMT + Placebo; Test type: Superiority; p = 0.15, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected through Week 26 (6 months).
Arm/Group | FMT + Bezlo | FMT + Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 5/30 | 4/31
Other Adverse Events (participants affected / at risk) | 16/30 | 15/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FMT + Bezlo (N=30) | FMT + Placebo (N=31)
IBD Flare (Gastrointestinal disorders) | 0 (0) | 1 (1) — Subject was hospitalized due to a UC flare, the study team determined it not to be related to FMT procedure. The adverse event resolved, and the subject continued in the study.
IBD Flare (Gastrointestinal disorders) | 0 (0) | 1 (1) — Subject was hospitalized due to a UC flare causing abdominal pain, the subject was discontinued from the trial prior to receiving study drug.
Colectomy (Gastrointestinal disorders) | 1 (1) | 0 (0) — Subject was admitted due to IBD complications, and surgical laparoscopy with complete colectomy and ileostomy by abdominal approach was performed. Post-op was uncomplicated, and subject was discharged.
IBD Flare (Gastrointestinal disorders) | 1 (1) | 0 (0) — Subject was admitted to the hospital for increased abdominal pain due to an IBD flare, the adverse event was resolved. The IBD flare occurred prior to administration of study drug, the subject continued in the study with no further issues.
Hospitalization (Gastrointestinal disorders) | 0 (0) | 1 (1) — Subject was hospitalized for worsening of ongoing baseline symptoms of rectal bleeding, diarrhea, and abdominal pain. The patient was treated for these symptoms and this adverse event was resolved.
IBD flare (Gastrointestinal disorders) | 0 (0) | 1 (1) — Subject experienced an IBD flare for which they were hospitalized. Patient was started on biologic treatment and deemed clinically stable for discharge.
IBD flare (Gastrointestinal disorders) | 1 (1) | 0 (0) — Subject experienced flare symptoms, which was treated by switching their IBD medications. The patient's symptoms improved with the treatment.
Colectomy (Gastrointestinal disorders) | 1 (1) | 0 (0) — Subject was admitted to the hospital for pain and nausea. They underwent total abdominal colectomy and end ileostomy and were discharged with antibiotics.
Hospitalization (Gastrointestinal disorders) | 1 (1) | 0 (0) — Subject was admitted for abdominal pain, diarrhea, and vomiting. They received IV steroids and antibiotics prior to discharged which resolved symptoms.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FMT + Bezlo (N=30) | FMT + Placebo (N=31)
Diarrhea (Gastrointestinal disorders) | 8 | 7
Rectal Bleeding (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 7 | 6
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Chest Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Fatigue (General disorders) | 2 | 1
Headache (General disorders) | 1 | 1
Fever (General disorders) | 1 | 1
Fecal urgency (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Dermatitis Radiation (Injury, poisoning and procedural complications) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Herpes Simplex Reactivation (Infections and infestations) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Bloating (Gastrointestinal disorders) | 0 | 1
Allergic reaction (Immune system disorders) | 1 | 0
Thrombocytopenia (Vascular disorders) | 0 | 1
COVID-19 Infection (General disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This study was limited by the sample size as well as the inclusion of PCR only testing for the qualifying episode. .

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT03829475/Prot_SAP_000.pdf